CLINICAL TRIAL: NCT06620523
Title: Efficacy of Mitochondrial Directed Therapy in Prevention of Cardiac Surgery Associated AKI Prevent Cardiac Surgery Associated AKI Trial (Prevent CSA-AKI Trial)
Brief Title: Prevent Cardiac Surgery Associated AKI Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, yoosif abdalla, Principal Investigator, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCR224635
Record Dates: First submitted 2024-07-30; First posted 2024-10-01 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Renal Failure; Coronary Artery Disease; Surgery; Surgery-Complications
Keywords: cardiac surgery; critical care medicine; anesthesiology; nephrology; cardiopulmonary bypass; renal failure; aki; supplement
MeSH Terms: conditions — Renal Insufficiency; Coronary Artery Disease | interventions — coenzyme Q10; Glutathione

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinded: study team, including principal investigator, sub-investigators, study coordinators, hospital pharmacy and medical students. Patient is also blinded.
  Unblinded: investigational drug pharmacists, investigational drug pharmacy technicians, nurses administering medication
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: CoQ10 1200 mg orally with Glutathione 1000 mg orally (Active Comparator): White-colored CoQ10 400 mg capsules will be dispensed AND White colored L-Glutathione 500 mg capsules will be dispensed.
  Interventions: Drug: CoQ10 1200 mg orally with Glutathione 1000 mg orally
- Group B: Placebo CoQ10 orally and Placebo Glutathione orally (Placebo Comparator): A placebo to exactly match the CoQ10 will be made with white gelatin empty capsules containing cellulose AND a placebo to exactly match the L-Glutathione will be made with white gelatin empty capsules containing cellulose.
  Interventions: Drug: Group B: Placebo CoQ10 orally and Placebo Glutathione orally

INTERVENTIONS:
Drug: CoQ10 1200 mg orally with Glutathione 1000 mg orally — This is the intervention to assess efficacy of CoQ10 and Glutathione in prevention of cardiac surgery associated acute kidney injury
  Arms: Group A: CoQ10 1200 mg orally with Glutathione 1000 mg orally
Drug: Group B: Placebo CoQ10 orally and Placebo Glutathione orally — A placebo to exactly match the CoQ10 will be made with white gelatin empty capsules containing cellulose AND a placebo to exactly match the L-Glutathione will be made with white gelatin empty capsules containing cellulose.
  Arms: Group B: Placebo CoQ10 orally and Placebo Glutathione orally

SUMMARY:
Prevent CSA-AKI (Cardiac Surgery Associated Acute Kidney Injury) trial is a double blinded randomized controlled trial, 242 patients undergoing elective cardiopulmonary bypass surgery (CPB)will either receive a placebo or daily 1200 mg of Co enzyme Q10 (CoQ10) and 1000 mg of Glutathione (GSH), the first dose will be given the day before surgery and continues while admitted up to 1 week. Blood and urine samples will be collected. Adverse events related to the study drugs will be collected.

DETAILED DESCRIPTION:
AKI (Acute Kidney Injury) is a serious and common complication post Cardiac surgery requiring cardiopulmonary bypass (CPB), the incidence is up to 30% Independent predictor for 30-day mortality, with a 41 % & % 62% in AKI stage III without and with the needs for RRT (Renal Replacement Therapy) respectively It's also associated with an a 3-fold increase in the long-term risk of ESRD (End Stage Renal Disease) Despite the high burden of CPB-induced AKI, our understanding of the pathophysiology still primitive, that makes us limited in designing directed therapies for prophylaxis, early detection and interventions that can lower its incidence, severity and progression. CPB induced AKI is multifactorial, however, renal ischemia-reperfusion injury (RIRI) is considered a major factor, poor renal perfusion driven by hemodynamic and volume changes, increased systemic inflammation, endothelial and epithelial cell injury and perioperative use of nephrotoxic agents all contribute to AKI post cardiac surgery.

Renal mitochondrial dysfunction has been implicated in the pathogenesis of RIRI, reperfusion following ischemia causes opening of mitochondrial permeability transition pore (MPTP), leading to depolarization of mitochondrial membrane, increased production of reactive oxygen species (ROS) and release of apoptotic proteins mitochondrial disruption contributes to impairment of ATP dependent cellular repair mechanisms, cell death, and persistent suppression of mitochondrial biogenesis, a process of which cells form new mitochondria furthermore, cell injury releases mitochondrial endogenous damage associated molecular patterns (DAMPs), Mitochondrial DAMPs (MTD) activates toll-like receptor-9 (TLR9) which results in innate immune cascade activation and further renal injury Loss of Mitochondrial function and integrity has been linked to initiation, progression and recovery phases of ischemia/ reperfusion acute kidney injury. In mice subjected to Sham surgery, UmtDNA (Urinary Mitochondrial Deoxyribonucleic Acid) increased after 10 min of ischemia, positively correlated with ischemia time and negatively correlated with renal cortical mtDNA and mitochondrial gene expression Levels of UmtDNA in AKI was evaluated with different population and different results. UmtDNA level correlated with renal function recovery but not with AKI severity following cardiac surgery. Same finding of correlation between UmtDNA with renal recovery was observed but wasn't statistically significant, additionally UmtDNA level reflected the severity of AKI and duration of renal replacement therapy in patients admitted with AKI Co Q10 or ubiquinone is an essential mitochondrial co-factor that has a critical role as a component of the electron transport chain and free radical scavenger. Co Q10 levels were found to be low in critically ill patients, lower levels found in post cardiac arrest with correlation poor neurological outcome and higher mortality. American heart association included CoQ10 as a promising neuroprotective agent, significantly lower left ventricular ejection fractions (LVEFs) seen in the lowest tertile of CoQ10 Biopsies taken from patients with cardiomyopathy showing increasing severity of heart disease correlate with lower levels of serum and myocardial deficiency of CoQ10, supplementation with CoQ10 resulted in significant increases in both myocardial and serum levels as well as reduction of disease severity. Coenzyme Q10 as Adjunctive Treatment of Chronic Heart Failure has shown that CoQ10 supplement reduced the primary 2-year end point of cardiovascular death, hospital stays for HF (Heart Failure), or mechanical support or cardiac transplant. It was also demonstrated that CoQ10 reduced the risk of congestive heart failure hospitalization and its complications like pulmonary edema and cardiac asthma Q12 supplement is safe and widely available as an over-the-counter, CoQ10 is available as ubiquinol (reduced form) or ubiquinone (oxidized form), Additionally, the ubiquinol containing formulation resulted in a higher plasma CoQ10 levels compared with ubiquinone formulations after a single dose of supplement. Dose of 1200 mg chose based on safety shown in many clinical trial data for CoQ10. The half-life of CoQ10 is 21.7 h (28 Mitochondria consume about 90% of the cellular O2 for ATP (Adenosine Tri-Phosphate) synthesis through oxidative phosphorylation, optimizing mitochondrial function and reducing oxygen free radicals may enhance cellular function and mitigate cellular injury thereby leading to improved outcome. Despite the accumulating evidence on the relevance of mitochondrial dysfunction in AKI initiation and progression and the crucial role mitochondrial therapies such as Co Q10 & Glutathione would play in renal protection and recovery, human data in this field are very limited. Using renal scintigraphy & immunohistochemical evaluation, it was demonstrated that CoQ10 decreased tissue oxidative stress levels, scores of histopathology and apoptosis; and decreased quantitative scintigraphic parameters with increased split renal function in ischemic kidney. The mitochondria-targeted Triphenylphosphine CoQ10 nanoparticles (T-NPCoQ10) which resulted in alleviation of mtDNA damage, suppressed inflammatory and apoptotic responses, and improved renal function in both cell and animal models. In human Co Q10 with Trimetazidine significantly lowered the incidence of Contrast induced nephropathy in previous research.

Glutathione (GSH): In addition to Oxidative stress as a key in cardiac surgery associated AKI; iron-dependent lipid peroxidation resulting in cell death play an important role, this process starts with intracellular glutathione (GSH) depletion. Glutathione S-transferases (GST) are a diverse group of phase II detoxification enzymes that works as a scavenger through conjugation of glutathione to a wide variety of electrophiles and reactive oxygen species. Alpha-GST isoform(a-GST) has specificity for the proximal tubule, and pi- GST isoform(pi-GST) that's confined to distal tubule.

It was demonstrated that post cardiac surgery Urinary pi- GST levels predicted development of AKI and overall prognosis in ischemia/reperfusion mouse models that total GST activity is reduced by ~35% during (0 4 h) AKI "initiation" and (18 or 72 h) "maintenance" phases. In previous research, acute kidney injury model established by systemic glutathione depletion in mice. In patients undergoing cardiac surgery, low levels of cardiac and systemic glutathione found to correlate to the functional status and structural cardiac abnormalities of patients with cardiac diseases it was shown that that high levels of serum GST Pi in the first 6 h after birth are associated with an increased AKI and mortality in prematurely born neonates. Experiment showed exogenous glutathione supplement alleviated Gentamicin induced AKI in rats intoxicated with gentamycin, partially by inhibiting oxidative stress, and intrinsic apoptosis. Glutathione supplements are safe and already available over the counter, studies have shown effectiveness of daily Glutathione administration at elevating stores of Glutathione and impacting the immune function and levels of oxidative stress

ELIGIBILITY:
Inclusion Criteria:

* Adult 18-70 years of age
* Undergoing elective CPB (Cardiopulmonary Bypass) surgery
* Baseline GFR (Glomerular Filtration Rate) ≥45 ml/min

Exclusion Criteria:

* GFR (Glomerular Filtration Rate) <45 ml/min
* Solitary kidney
* Status post-kidney transplant
* Pregnant women
* Allergy to CoQ10
* Allergy to Glutathione
* Allergy to Cellulose

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2027-06-17 (Estimated); Study Completion 2028-06-17 (Estimated)

PRIMARY OUTCOMES:
AKI incidence reduction | 28 days
  Reduction of cardiac surgery associated acute kidney injury
AKI incidence reduction | 90 days
  Reduction of cardiac surgery associated acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: Yoosif Abdalla, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States

DOCUMENTS (4):
  • Study Protocol (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT06620523/Prot_000.pdf
  • Statistical Analysis Plan: Data definitions (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT06620523/SAP_001.pdf
  • Statistical Analysis Plan: Data definitions (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT06620523/SAP_002.pdf
  • Informed Consent Form (2024-09-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT06620523/ICF_003.pdf